CLINICAL TRIAL: NCT06922851
Title: Protein A Immunoadsorption in Dilated Cardiomyopathy: A Prospective, Multicenter, Randomized Study to Evaluate Efficacy and Safety (PRIA-DCM)
Brief Title: Protein A Immunoadsorption in Dilated Cardiomyopathy (RPIA-DCM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRIA-DCM
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Dilated Cardiomyopathy (DCM)
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Plasmapheresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immuoadsorption group (Experimental): receiving immunoadsorption therapy
  Interventions: Procedure: Immunoadsorption
- Control group (No Intervention): not receiving immunoadsorption therapy

INTERVENTIONS:
Procedure: Immunoadsorption — Immunoadsorption (IA) therapy using a protein A column for four consecutive days, plus immunoglobulin supplementation after IA
  Arms: Immuoadsorption group

SUMMARY:
This study is a multicenter, dual-arm and randomized controlled clinical trial. Sixty patients with dilated cardiomyopathy and positive β1-adrenergic receptor autoantibodies were selected and randomly divided into an immunoadsorption group (receiving immunoadsorption therapy) and a control group in a 1:1 ratio. Changes in cardiac function, morphology and clinical outcomes were followed up and compared.

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy
* Presence of anti-β1-adrenergic receptor
* Age 18-75 years
* LVEF ≤ 40% determined by echocardiography (according to assessment of the local investigators)
* NYHA class II-IV
* Symptoms of heart failure ≥ 6 months
* Treatment with guideline-directed medical therapy (GDMT) for ≥6 months and stable dose of ACEI/ARB/ARNI/β-blocker/SGLT2i/MRA/sGCa for ≥1 month (excluding diuretics)
* Hemodynamically stable
* Informed consent

Exclusion Criteria:

* ICD implantation < 1 month or CRT/D implantation < 6 months
* Heart failure caused by other heart diseases
* End-stage heart failure, inability to discontinue intravenously positive inotropic or vasoactive drugs
* Expected survival < 1 year
* Hemoglobin < 90g/L
* Any disease requiring immunosuppressive drugs
* Commodities with other acute or severe illnesses, such as infections, severe hepatic or renal dysfunction, hematological diseases, malignant tumors, cachexia, autoimmune diseases, etc.
* Previous treatment with immunoadsorption therapy or intravenous immunoglobulin therapy
* Contraindications to extracorporeal circulation therapy, such as mental illness or consciousness disorders, shock, severe bleeding or bleeding tendency, coagulation dysfunction, multiple organ failure, etc.
* Pregnancy/lactation
* Any other conditions that the researcher deems may increase the risk to the subject or interfere with the clinical trial and outcome assessment (such as excessive anxiety, alcohol or drug abuse, or cognitive impairment, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-04 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in LVEF from baseline to 6 months determined by echocardiography | From enrollment to follow-up at 6 months

SECONDARY OUTCOMES:
LVEF as determined by echocardiography at baseline and after 3, 12 and 24 months | From enrollment to follow-up at 24 months
LVEDD and LVESD as determined by echocardiography at baseline and after 3, 6, 12 and 24 months | From enrollment to follow-up at 24 months
NYHA classification at baseline and after 3, 6, 12 and 24 months | From enrollment to follow-up at 24 months
Kansas City Cardiomyopathy Questionnaire (KCCQ) score at baseline and after 3, 6, 12 and 24 months | From enrollment to follow-up at 24 months
  KCCQ score is scaled from 0 to 100 and higher scores mean better health status.
NT-proBNP at baseline and after 3, 6, 12 and 24 months | From enrollment to follow-up at 24 months

OTHER OUTCOMES:
Safety outcome | From enrollment to follow-up at 24 months
  The occurrence of adverse events (AE) and serious adverse events (SAE)
Exploratory outcome and analyses | From enrollment to follow-up at 24 months
  Composite of all-cause mortality, heart transplantation, implantation of LVAD or hospitalization for heart failure at 24 months; Symptom duration; Genetic variants; Serum levels of IgG, IgA, IgM, IgD, IgE and IgG subclasses at baseline, treatment day 1 to 4 (twice every day: before treatment and within 1 h after treatment), day 5 and month 3, 6, 12 and 24; Serum levels of anti-β1-adrenergic receptor at baseline, day 5, months 3, 6, 12 and 24; Serum levels of autoantibodies at baseline and after 3, 6, 12 and 24 months; Cardiac structure, function and fibrosis assessed using cardiac magnetic resonance imaging at baseline and 6-month.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Cheng, M.D., Ph.D., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No